CLINICAL TRIAL: NCT07257159
Title: End-of-Life Care Preparedness Program for Senior Nursing Students: Effects on Attitudes and Self-Efficacy in a Randomized Controlled Trial
Brief Title: End-of-Life Care Preparedness Program for Senior Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hilal ALTUNDAL DURU (Other)
Responsible Party: Sponsor-Investigator, Hilal ALTUNDAL DURU, Doctor, Mersin University
Organization: Mersin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KaratekinU
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Self-Efficacy; Attitude; End-of-Life Care
Keywords: Death education; End-Of-Life; Nursing students; Self-efficacy
MeSH Terms: conditions — Behavior; Death

STUDY DESIGN:
Intervention Model Description: The study was planned as a prospective (pre-post-fallow up test), two-armed (1:1), randomized controlled experimental study. This randomized controlled trial will be reported according to the CONSORT guidelines.
Who Masked: Participant
Masking Description: Senior nursing students in the intervention and control groups will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The End-of-Life Care Preparedness Program will be held in a online environment for the students in the intervention group. This training program has been developed based on the literature. The primary aim of the program was to enable participants to recognize their own thoughts and emotions about death, and to support their development in key areas of end-of-life care. Specifically, the content addressed providing care to dying individuals, caring for the deceased person, preparing the body after death, and offering psychosocial support to the bereaved family. The intervention consisted of four weekly sessions, each lasting approximately 90 minutes, delivered in an online group format via online. The training program will be applied to 29 senior nursing students in the intervention group. The sessions were structured to include psychoeducational content, interactive exercises, group discussions, and opportunities for reflection.
  Interventions: Other: The End-of-Life Care Preparedness Program
- Control (No Intervention): There will be no training or intervention.

INTERVENTIONS:
Other: The End-of-Life Care Preparedness Program — The End-of-Life Care Preparedness Program will be held in a online environment for the students in the intervention group. This training program has been developed based on the literature. The primary aim of the program was to enable participants to recognize their own thoughts and emotions about death, and to support their development in key areas of end-of-life care. Specifically, the content addressed providing care to dying individuals, caring for the deceased person, preparing the body after death, and offering psychosocial support to the bereaved family. The intervention consisted of four weekly sessions, each lasting approximately 90 minutes, delivered in an online group format via online. The training program will be applied to 29 senior nursing students in the intervention group. The sessions were structured to include psychoeducational content, interactive exercises, group discussions, and opportunities for reflection.
  Arms: Intervention

SUMMARY:
In this study, between 1 April- 31 May 2025, who met the inclusion and exclusion criteria, a total of 59 senior nursing students who are with 4th year nursing students starting the Nursing Department of Çankırı Karatekin University and Sakarya Applied Sciences University.

DETAILED DESCRIPTION:
The End-of-Life Care Preparedness Program will be held in a online environment for the students in the intervention group. This training program has been developed based on the literature. The primary aim of the program was to enable participants to recognize their own thoughts and emotions about death, and to support their development in key areas of end-of-life care. Specifically, the content addressed providing care to dying individuals, caring for the deceased person, preparing the body after death, and offering psychosocial support to the bereaved family. The intervention consisted of four weekly sessions, each lasting approximately 90 minutes, delivered in an online group format via online. The training program will be applied to 29 senior nursing students in the intervention group. The sessions were structured to include psychoeducational content, interactive exercises, group discussions, and opportunities for reflection.

ELIGIBILITY:
Inclusion Criteria:

* final-year nursing students
* consent to take part voluntarily
* accessed to the required technology and competencies for attending online sessions

Exclusion Criteria:

* failed to complete the data collection tools in full
* missed intervention sessions
* chosed to withdraw at any point during the intervention or follow-up phase

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
End-of-Life and Postmortem Self-Efficacy Scale (ELPSES) | Change from before education (Time 0) and after education (four weeks-Time 1) up to after the at the end of the education one month later (Time 2).
  This instrument was evaluate nursing students' self-efficacy regarding end-of-life and postmortem care. The scale consists of 18 items and is formatted as a visual analog scale. For each item, participants indicate their perceived level of self-efficacy on a continuum from 0 (not confident at all) to 100 (extremely confident) using a slider mechanism. The overall self-efficacy score is calculated by averaging responses across items. In the original development study, the Cronbach's alpha for the scale was reported as 0.93.
Frommelt Attitudes Toward Care of the Dying Scale (FATCOD) | Change from before education (Time 0) and after education (four weeks-Time 1) up to after the at the end of the education one month later (Time 2).
  The FATCOD, originally developed by Frommelt (1991), was used to assess participants' attitudes toward caring for dying patients. The Turkish adaptation and validation of the scale was conducted by Çevik and Kav (2013). The scale contains 30 items rated on a 5-point Likert scale and includes both positively and negatively worded statements. Negative items are reverse-coded before computing the total score, which ranges from 30 to 150, with higher scores indicating more positive attitudes toward caring for dying patients. In the Turkish validation study, the Cronbach's alpha reliability coefficient was reported as 0.73.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal ALTUNDAL DURU, PhD, Principal Investigator — Çankırı Karatekin University
Locations (1):
- Çankırı Karatekin University, Çankırı, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No